CLINICAL TRIAL: NCT01036724
Title: Comparative Study of Guided Radiofrequency Ablation Using the CARTO® 3 and NavX™ Systems for the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: Guided Radiofrequency Ablation Using the CARTO® 3 and NavX™ Systems for the Treatment of Paroxysmal Atrial Fibrillation
Acronym: CO1
Status: Terminated | Type: Observational
Why Stopped: Enrollment challenges
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BWICO1
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-08

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Carto 3: Those subjects whose cases use the CARTO 3 EP Navigation System.
  Interventions: Device: Cardiac Mapping
- NAVX: Those subjects whose cases use the NAVX(TM) EP Navigational System.
  Interventions: Device: Cardiac Mapping

INTERVENTIONS:
Device: Cardiac Mapping — Generating a cardiac map using the study device (CARTO 3) compared to the control device (NAVX[TM]) and measuring the amount of radiation exposure duration for each.

SUMMARY:
The purpose of this study is to determine the change in median radiation exposure time and median procedure time following guided radiofrequency (RF) ablation among subjects undergoing treatment for paroxysmal atrial fibrillation with either the CARTO® 3 or the NavX(TM) System.

It is hypothesized that described features will reduce the median radiation exposure during the CARTO® 3 system-guided procedures compared to the NavX(TM) system-guided procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for a first radiofrequency ablation procedure for treatment of paroxysmal atrial fibrillation (AF episodes that last less than 30 days and are not terminated via cardioversion) and who are considered eligible for treatment by the physician.

Exclusion Criteria:

* There are no study specific exclusion criteria for this observational study. The exclusion criteria will be conditions that, in the physicians opinion, preclude an RF ablation procedure because the procedure risks outweigh any potential benefits for the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred for Radiofrequency ablation treatment for paroxysmal atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2010-08-01 (Actual); Study Completion 2010-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Vancouver Island Health Authority - Royal Jubilee Hospital, Victoria, British Columbia
  - QE II Health Sciences Center, Halifax, Nova Scotia
  - London Health Sciences, London, Ontario
  - Southlake Regional Healthcare Centre, Newmarket, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Laval Hopital, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carto 3 | NAVX
Started | 52 | 55
Completed | 46 | 47
Not Completed | 6 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carto 3 | NAVX | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Median (Full Range); unit: years] | 58 [22 to 74] | 57 [36 to 79] | 58 [22 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 32 | 40 | 72

OUTCOME MEASURES:

1. Primary Outcome: Total Fluoroscopy Time
Description: The primary outcome measure of this study is to measure and compare total fluoroscopy exposure time (minutes) at the conclusion of radiofrequency ablation for the treatment of paroxysmal atrial fibrillation, when guided by the CARTO® 3 or the NavX(TM) System in similar procedures.
Time Frame: Throughout the Total Duration of the Procedure
Measure: Median (Full Range); unit: minutes
Arm/Group | Carto 3 | NAVX
Number analyzed (Participants) | 46 | 47
minutes | 31.0 [0.7 to 61.6] | 37.5 [4.3 to 76.0]

2. Secondary Outcome: Total Procedure Time
Time Frame: Total Duration of the Procedure
Measure: Median (Full Range); unit: minutes
Arm/Group | Carto 3 | NAVX
Number analyzed (Participants) | 46 | 47
minutes | 160.5 [82.0 to 414.0] | 147.0 [86.0 to 343.0]

ADVERSE EVENTS:
Time Frame: Throughout the Duration of the Procedure
Arm/Group | Carto 3 | NAVX
Serious Adverse Events (participants affected / at risk) | 1/46 | 3/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carto 3 (N=46) | NAVX (N=47)
Atrial Perforation (Cardiac disorders) | 0 (0) | 2 (2) — Not related to imaging technology
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 1 (1) — Not related to imaging technology

LIMITATIONS AND CAVEATS:
The study was terminated early, with 107 enrolled and 93 evaluable subjects, due to difficulty enrolling despite prolonged extension of the enrollment period. The original design called for 176 enrolled and 122 evaluable patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No